CLINICAL TRIAL: NCT06132997
Title: Medical Thoracoscopy Versus Conventional Intercostal Tube in Treatment Outcomes of Empyema Management
Brief Title: Medical Thoracoscopy in Treatment Outcomes of Empyema Management
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hend Mohamed Sayed Mohamed (Other)
Responsible Party: Sponsor-Investigator, Hend Mohamed Sayed Mohamed, Principal investigator, Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Medical thoracoscopy&Empyem
Record Dates: First submitted 2023-10-26; First posted 2023-11-15 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Empyema
MeSH Terms: conditions — Empyema

STUDY DESIGN:
Intervention Model Description: Medical thoracoscopy group
Who Masked: Participant
Masking Description: Intercostal chest tube group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medical thoracoscopy group (Active Comparator): Medical thoracoscopy is a minimally invasive endoscopic procedure utilized by pulmonologists to evaluate, diagnose, and treat pleural pathologies of the lung, mainly pleural effusions.
  Interventions: Procedure: Thoracoscopy procedure; Procedure: Chest tube thoracostomy
- Intercostal tube group (Active Comparator): Intercostal chest tube placed without thoracoscopy for patients with confirmed empyema.
  Interventions: Procedure: Thoracoscopy procedure; Procedure: Chest tube thoracostomy

INTERVENTIONS:
Procedure: Thoracoscopy procedure — is a minimally invasive endoscopic procedure utilized by pulmonologists to evaluate, diagnose, and treat pleural pathologies of the lung, mainly pleural effusions.
Procedure: Chest tube thoracostomy — Insert chest intercostal tube without thoracoscopy

SUMMARY:
To evaluate the efficacy of drainage achieved by thoracoscopy vs tube drainage alone.

To compare clinical outcomes such as length of hospital stay, need for additional procedures, and treatment failure rates between the two drainage methods.

To asses resolution of pleural infection and rates of fluid re-accumulation over follow-up.

To compare safety profiles and complication rates of thoracoscopy versus tube drainage alone

DETAILED DESCRIPTION:
Empyema is a serious infection characterized by pus accumulation in the pleural space. Effective drainage and treatment is necessary for resolution. Traditionally, intercostal tube placement was standard initial management. However, recent studies have compared outcomes of early medical thoracoscopy or video-assisted thoracoscopic surgery (VATS).

Thoracoscopy enables direct visualization for thorough pleural space cleansing and debridement under direct vision. medical thoracoscopy significantly improved drainage adequacy and reduced treatment failure risks compared to tube drainage alone. Also reported shorter hospital stays and lower complication rates with early thoracoscopy-directed management.

Additional benefits of thoracoscopy include enabling talc pleurodesis for reducing empyema recurrence. thoracoscopy-directed pleurodesis achieved higher long-term success rates than tube drainage followed by pleurodesis. Overall, current evidence indicates medical thoracoscopy provides superior empyema treatment outcomes to conventional tube drainage through optimized drainage and debridement under direct visualization.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of empyema via Imaging tests (e.g. chest x-ray/CT scan)
* Age 18 years or older
* Clinical signs/symptoms consistent with Empyema such as fever, chest pain, coughs
* Pleural fluid loculations/septations seen on Imaging requiring drainage
* No previous drainage procedures done for Current empyema

Exclusion Criteria:

* Age less than 18 years
* Immunocompromised state or other conditions Contraindications to thoracoscopy
* Previous drainage procedure for current Empyema
* Residual pleural fluid not amenable to drain

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-12-24 (Estimated); Primary Completion 2024-12-28 (Estimated); Study Completion 2025-03-24 (Estimated)

PRIMARY OUTCOMES:
Treatment success: | baseline
  Asses by chest ultrasound

SECONDARY OUTCOMES:
Success of pleurodesis | baseline
  measured by assessing the recurrence rate of pleural effusion over a specified follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Ahmed, MD, Study Chair — Doctor

REFERENCES:
- [Background] Godfrey MS, Bramley KT, Detterbeck F. Medical and Surgical Management of Empyema. Semin Respir Crit Care Med. 2019 Jun;40(3):361-374. doi: 10.1055/s-0039-1694699. Epub 2019 Sep 16. PMID 31525811
- [Background] Aboudara M, Maldonado F. Update in the Management of Pleural Effusions. Med Clin North Am. 2019 May;103(3):475-485. doi: 10.1016/j.mcna.2018.12.007. PMID 30955515